CLINICAL TRIAL: NCT01942564
Title: The Head Injury-associated Photosensitivity and Pupillary Function (HIPP) Study
Acronym: HIPP
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Principal Investigator, Andrew Hartwick, Assistant Professor, Ohio State University
Other Study IDs: 2013H0151; W81XWH-12-1-0434 (Other Grant/Funding Number: Telemedicine and Advanced Technology Research Center)
Record Dates: First submitted 2013-09-06; First posted 2013-09-16 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Head Injury; Traumatic Brain Injury (TBI); Photosensitivity; Photophobia
Keywords: traumatic brain injury; photophobia; photosensitivity; pupil
MeSH Terms: conditions — Craniocerebral Trauma; Brain Injuries, Traumatic; Photosensitivity Disorders; Photophobia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Case Subjects: 1. Age 18 years or older
  2. Had a head injury that occurred at least 6 months prior to entering study
  3. Have found lights more bothersome since injury
- Control Subjects: 1. Age 18 years or older
  2. Have not had a previous head injury
  3. Have had a full eye examination at Ohio State University College of Optometry during last 6 months.

SUMMARY:
After a head injury, many people find that exposure to light causes them increased discomfort. By measuring how the pupil in the eye constricts to flashes of red and blue light, this study will investigate whether this phenomenon is due to a change in the eye's sensitivity to light.

DETAILED DESCRIPTION:
The pupils inside the eyes constrict in response to light stimulation. Different classes of cells within the human retina initiate this response. Recent research suggests that one of the ganglion cell types involved in this pupil response also plays a role in the photophobia experienced by migraine sufferers. The main aim of this study is to determine whether this type of ganglion cell becomes 'hypersensitive' after traumatic brain injury, thereby contributing to symptoms of increased photosensitivity experienced by many of these individuals.

In the first session of this study, subjects will be asked questions about their sensitivity to light and the reaction of their eyes' pupils to flashing red and blue lights will be measured. The subjects will be given a full eye examination to rule out other causes of increased photosensitivity.

In some cases, subjects will be asked to attend a second session roughly two weeks later. They will be asked to wear a watch that measures their daily activity/sleep rhythms and light exposure during this inter-session period. During the second session, further testing of the pupil responses to blue and red flickering light will be performed.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years old
* reports a previous head injury that occurred at least 6 months ago
* score of 2 or 3 (mild TBI) on OSU-TBI ID Survey
* best-corrected visual acuity of at least 20/30 in both eyes
* reliable visual field

Exclusion Criteria:

* pregnancy
* significant afferent pupillary defect
* previous history of neurodegenerative disease
* intraocular pressure more than 21 mm Hg
* significant visual field defect
* active corneal pathology
* history of retinal or optic nerve disease
* strabismus (eye turn)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cases: Age 18 or older with symptoms of increased photosensitivity since experiencing a head injury.
  Controls: Matched to cases in age, sex and race.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2013-08; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Pupil Responses | 2 weeks
  The pupil fluctuation evoked by blue and red flickering lights will be measured in patients with a prior brain injury and compared to matched controls.

SECONDARY OUTCOMES:
Sleep Rhythms | 2 weeks
  Daily rhythms of sleep and activity will be assessed in subjects with prior brain injury and compared to matched controls.
Light Exposure | 2 weeks
  The exposure to red, blue and green components of the light spectrum will be quantified in patients with a prior brain injury, and compared to matched controls.
Photosensitivity Symptoms | Single visit - one day
  Subjects will complete survey indicating symptoms they have experienced related to light sensitivity and will grade their discomfort after exposed to brief flashes of light.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Hartwick, OD, PhD, Principal Investigator — Ohio State University
Locations (1):
- College of Optometry, Columbus, Ohio, United States

REFERENCES:
- [Background] Barker F, Cockerham G, Goodrich G, Hartwick A, Kardon R, Mick AB, Swanson M. Brain Injury Impact on the Eye and Vision. Optom Vis Sci. 2017 Jan;94(1):4-6. doi: 10.1097/OPX.0000000000001001. No abstract available. PMID 28009763
- [Result] Yuhas PT, Shorter PD, McDaniel CE, Earley MJ, Hartwick AT. Blue and Red Light-Evoked Pupil Responses in Photophobic Subjects with TBI. Optom Vis Sci. 2017 Jan;94(1):108-117. doi: 10.1097/OPX.0000000000000934. PMID 27464575